CLINICAL TRIAL: NCT05082090
Title: A Multi-Center Post-Market Data Collection Protocol to Evaluate the Performance of Orthofix Spine Devices
Acronym: RWE Spine
Status: Active, not recruiting | Type: Observational
Sponsor: Orthofix Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-2001SPPM
Record Dates: First submitted 2021-09-21; First posted 2021-10-18 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Spinal Disorders/Injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Implanted with Orthofix Spinal products: Study will include 2000+ subjects implanted with Orthofix Spine devices including spine fixation systems and motion preservation systems (i.e. M6-C artificial cervical disc and M6-L artificial lumbar disc)
  Interventions: Procedure: Spinal Surgery

INTERVENTIONS:
Procedure: Spinal Surgery — Implanted with Orthofix Spinal products

SUMMARY:
This protocol is designed to study Orthofix regulatory approved and commercially available spine devices to generate Real World Evidence (RWE) of device safety and performance in the treatment of patients with spine injuries and/or disorders following the local medical standard of care. The clinical data generated from this study will support compliance to global regulatory requirements including but not limited to the European Medical Device Regulation (EU MDR) for the applicable devices.

ELIGIBILITY:
Inclusion Criteria:

1. Patient diagnosed with a spine injury/disorder and undergoing or has undergone spine procedure at the participating investigative centers utilizing Orthofix Spine devices.
2. Patient is 18 years or older at the time of surgery.
3. Patient is capable of understanding the content of the patient information / Informed Consent Form (ICF) for the prospective segment of the study.
4. Patient is willing and able to participate in the prospective data collection protocol and comply with the required data collection.

Note: For retrospective segment of the study: A waiver of consent for retrospective data collection is in place OR an informed consent is obtained from the participating patient prior to data collection as required by local regulations.

Exclusion criteria:

1. Patient may be excluded from study participation if there are other concurrent medical or other conditions (chronic or acute in nature) that in the opinion of the participating investigator may prevent participation or otherwise render patient ineligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Both retrospective and prospective study subjects have spinal injuries/disorders requiring treatment with an Orthofix Spine device.
  The three types of subject enrollment include:
  1. Retrospective data collection only
  2. Prospective data collection only
  3. Retrospective and prospective data collection
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Assessment: Device or procedure related adverse events | Pre-Operative to up to 10-years Post-Operative
  Evaluation of device related or procedure related adverse events
Primary Effectiveness Assessments: Fusion status measured radiographs | Intra-operative to up to 10-years Post-Operative
  Fusion status measured utilizing quantitative and qualitative radiographic assessments as applicable
Primary Effectiveness Assessment | Intra-operative to up to 10-years Post-Operative
  Improvement in pain measured with Visual Analogue Scale (VAS) or Numeric Rating Scale (NRS): NRS is an 11-point scale for patient self-reporting of pain. Patients rate their current pain intensity at the time of the visit from 0 ("no pain") to 10 ("worst possible pain") by selecting a number on a horizontal bar. NRS scores for the evaluation of pain have been categorized as mild (1-3), moderate (4-6), or severe (7-10). VAS scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
Primary Effectiveness Assessment | Intra-operative to up to 10-years Post-Operative
  Improvement in function as measured with Neck Disability Index (NDI) or Oswestry Disability Index (ODI).
  NDI includes 4 items that relate to subjective symptomatology (pain severity, headache, concentration, sleeping) and 6 items that relate to activities of daily living (lifting, work, driving, recreation, personal care, reading). Each item is scored from 0 to 5, with higher scores corresponding to greater disability. A total NDI score is determined by adding the scores of the individual questions and dividing that total by the maximum possible score (i.e., 50 if all questions are answered) to yield a percentage. Therefore, the NDI score ranges from 0 to 100. The ODI was developed as a specific outcomes tool for subjects suffering from back pain. The questionnaire scores 10 aspects of the subject's home and work life and analgesic use. The disability index is then calculated as a percentage with a high percentage indicating a high level of disability.

SECONDARY OUTCOMES:
Secondary Safety Assessments: Additional required medical treatments and/or supplemental surgical procedure | Pre-Operative to up to 10-years Post-Operative
  Additional required medical treatments and/or supplemental surgical procedure(s) at the index level (including revision, removal, reoperation, or supplemental fixation).
  Percentage of patients that required additional/supplemental treatments and/or surgical procedures and time to additional surgery.
Secondary Effectiveness Assessments: Quality of Life assessment | Pre-Operative to up to 10-years Post-Operative
  Quality of Life score measured utilizing PROMIS-29 PROMIS®-29 Profile v2. PROMIS (Patient-Reported Outcomes Measurement Information System) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. It can be used with the general population and with individuals living with chronic conditions. This instrument is comprised of 8 constructs: Physical Function; Anxiety; Depression; Fatigue; Sleep Disturbance; Ability to Participate in Social Roles and Activities; Pain Interference; and Pain Intensity that closely evaluate the impact of a patient's health on their quality of life
Secondary Effectiveness Assessments: Changes in neurological function | Pre-Operative to up to 10-years Post-Operative
  Maintenance or improvement in neurological function Neurological function will be evaluated, where neurological examination is performed as part of standard of care. The outcome of neurological function assessment (normal versus abnormal) and details related to abnormal sensory function (i.e. absent/impaired/normal/other) will be collected as appropriate.
Secondary Effectiveness Assessments: Work and Activity status | Pre-Operative to up to 10-years Post-Operative
  Work/Activity status
  Return to Work: The ability to and the time it takes for the subjects to return to work from the date of surgery will be documented.
  Return to Normal/Usual activities: The ability to and the time it takes for the subjects to return to normal daily activities from the date of surgery will be documented.
Secondary Effectiveness Assessments: Patient Satisfaction | Pre-Operative to up to 10-years Post-Operative
  Patient satisfaction At ≥ 6-months after the index procedure, subjects will be asked how satisfied they are with the results of their surgery on a 5-point Likert Scale (Very Satisfied; Satisfied; Neutral; Unsatisfied; Very Unsatisfied).
Secondary Effectiveness Assessments: Duration of Surgery | Pre-Operative to up to 10-years Post-Operative
  Surgery time
Secondary Effectiveness Assessments: Duration of Hospital stay | Pre-Operative to up to 10-years Post-Operative
  Length of hospital stay
Secondary Safety Assessments: Device and/or procedure-related deficiencies | Pre-Operative to up to 10-years Post-Operative
  Quantitative and qualitative radiographic assessments for evidence of device and/or procedure-related deficiencies.
  Inadequacy of a medical device with respect to its identity, quality, durability, reliability, usability, safety or performance will be documented. Percentage of patients with device deficiency will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Cahit Akbas, Study Director — Global Clinical Program Manager
Locations (20):
- United States (9):
  - Lanman Spinal Neurosurgery, Beverly Hills, California
  - RasouliSpine, Beverly Hills, California
  - Neurosurgical Medical Clinic, San Diego, California
  - Acadiana Neurosurgery, Lafayette, Louisiana
  - Columbus Orthopaedic, Columbus, Mississippi
  - M3 Emerging Medical Research, Durham, North Carolina
  - University Orthopedics, East Providence, Rhode Island
  - Summit Brain, Spine and Orthopedics, Lehi, Utah
  - Tuckahoe Orthopedics, Richmond, Virginia
- Germany (5):
  - Marien-Krankenhaus Bergisch Gladbach, Bergisch Gladbach
  - Stenum Ortho GmbH, Ganderkesee
  - Praxis für Neurochirurgie-Chirotherapie, Nordhausen
  - Orthopädikum Potsdam, Potsdam
  - Krankenhaus Maria-Hilf Stadtlohn, Stadtlohn
- South Africa (2):
  - The Club Surgical Centre, Pretoria
  - Zuid-Afrikaans Hospital, Pretoria
- Spain (4):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario Son Espases, Palma de Mallorca
  - University Hospital Marqués de Valdecilla, Santander

IPD SHARING:
Plan to Share IPD: No